CLINICAL TRIAL: NCT06957327
Title: A Phase 1b/2 Study of ERAS-601 SHP2 Inhibitor as a Monotherapy in Patients With Advanced and Progressing Chordoma
Brief Title: A Study of ERAS-601 in People With Chordoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-071
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Chordoma
Keywords: Advanced and Progressing Chordoma; ERAS-601 SHP2 Inhibitor; 25-071
MeSH Terms: conditions — Chordoma

STUDY DESIGN:
Intervention Model Description: The Phase 1b portion is a single-arm, single-center pilot study to evaluate the efficacy and safety of SHP2 inhibitor ERAS-601 for the treatment of advanced and progressing chordoma.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ERAS-601 (Experimental): All patients on the single-arm Phase 1b study will take ERAS-601 40mg BID, 3-weeks on 1-week off (3/1), as monotherapy. Each treatment cycle consists of a 4-week (28-day) treatment period.
  Interventions: Drug: ERAS-601

INTERVENTIONS:
Drug: ERAS-601 — ERAS-601 40mg BID, 3-weeks on 1-week off (3/1), as monotherapy

SUMMARY:
The researchers are doing this study is to find out whether ERAS-601 is a safe and effective treatment that causes few or mild side effects in people with advanced and progressing chordoma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Have histologically confirmed chordoma that is not dedifferentiated or poorly differentiated subtype.
* Have progressive disease per RECIST 1.1 defined by +20% change between any two scans in the 9 months prior to enrollment.
* Have Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 1
* Recovered from acute, clinically significant toxicities associated with current/recent treatments to acceptable baseline status
* Screening laboratory values must meet the following criteria and should be obtained within 30 days prior to study treatment:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 103/m
  * Platelet count ≥ 75 × 103/mL without symptomatic bleeding
  * Hemoglobin > 9 g/dL
  * Serum electrolytes (sodium, potassium, magnesium, phosphorus, calcium) Grade ≤1 or within the institutional ranges of normal. If clinically appropriate, electrolytes may be corrected, and values reassessed prior to enrollment.
  * AST and ALT ≤ 2.5 × ULN or ≤ 5 × ULN for patients with liver metastases
  * Total bilirubin ≤ 1.5 × ULN (except in patients with Gilbert Syndrome who can have total bilirubin < 3.0 mg/dL)
  * Serum creatinine clearance <1.5 times ULN or ≥ 50 mL/min as determined by Cockcroft-Gault (Appendix 7) (creatinine clearance need not be calculated if serum creatinine is within normal limits).

Female patients of childbearing potential must have a negative serum beta-human chorionic gonadotropin pregnancy test within 7 days prior to receiving the first dose of study medication.

* Female patients of childbearing potential must be willing to use an adequate method of contraception, as outlined in the protocol, for the course of the study through 120 days after last dose of study medication.
* Male patients of childbearing potential must agree to use an adequate method of contraception, as outlined in the protocol, starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Willing to comply with all protocol required- visits, assessments, and procedures.
* Willing to participate in patient interviews for quality-of-life assessment and complete patient reported outcomes (PRO) questionnaires
* Non-English speaking patients will not be required to complete patient reported outcomes.

Exclusion Criteria:

* Previous treatment with a SHP2 inhibitor.
* Documented PTPN11 mutations.
* Is currently receiving another treatment within 4 weeks of the first dose of ERAS-601 that may impact the outcome of this trial.
* Patients with prior antineoplastic therapy within <21 days or 5 half-lives, whichever is shorter.
* Received radiation within 14 days of Cycle 1, Day 1.
* Received strong inhibitors or inducers of CYP3A4, including grapefruit, grapefruit juice, and herbal supplements from 7 days prior to the administration of study drug.
* History of calcium and phosphate homeostasis disorder or systemic mineral imbalance with ectopic soft tissue calcification.
* Gastrointestinal dysfunction that may affect drug absorption.
* Have an untreated, uncontrolled, active infection (bacterial, fungal, or viral) requiring treatment that will impact this protocol.
* History or current evidence of retinal pigment epithelial detachment (RPED), central serous retinopathy, retinal vein occlusion (RVO), or predisposing factors to RPED or RVO.
* Sight-limiting degenerative corneal opacity.
* Have any underlying medical condition (e.g. cardiac, pulmonary, hepatic, etc.), psychiatric condition, or social situation that, in the opinion of the Investigator, would compromise patient safety and/or efficacy evaluation as per protocol.
* Incomplete recovery or ongoing complications from prior surgery that in the opinion of the principal investigator will compromise safety of patient and/or efficacy evaluation of protocol.
* Are pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of study therapy.
* Have a second malignancy that is active and in the opinion of the principal investigator will compromise safety of patient and/or efficacy evaluation of protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Clinical Benefit Rate (Phase Ib) | 1 year
  proportion of patients with CR or PR at any time or SD ≥ 6 months per RECIST 1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Mrinal Gounder, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center - Suffolk (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org